CLINICAL TRIAL: NCT05581953
Title: The Role of Lean-pork Within a Plant-based Dietary Pattern for Improving Iron Reserve, Muscle-fitness, and Markers of Health Span in Older Adults: A Multi-disciplinary Randomized Controlled Feeding Study
Brief Title: Protein-Distinct Macronutrient-Equivalent Diet 2
Acronym: PRODMED2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Principal Investigator, Moul Dey, Professor, South Dakota State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-2209010-EXP
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Blinding will be implemented to the extent possible. A researcher, unaware of the study goals and not involved with downstream data analyses will use a 1:1 block randomization to allocate participants to the diets in the first arm. Food service personnel (care provider) will not be aware of study goals and allocations. Metabolomic assays will be run in a blinded manner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-ultra-processed Omnivorous (Experimental): Minimally processed animal protein-lean pork within a low UPF dietary pattern
  Interventions: Other: Omnivorous
- Low-ultra-processed No meat (Other): Plant-forward no meat
  Interventions: Other: No meat

INTERVENTIONS:
Other: Omnivorous — Pork-added plant-forward diet
  Arms: Low-ultra-processed Omnivorous
Other: No meat — Plant-forward no meat
  Arms: Low-ultra-processed No meat

SUMMARY:
The central hypothesis is that the addition of minimally processed lean pork to a healthy plant-forward low ultra-processed diet will enhance nutrient adequacy, promote muscular fitness, and maintain metabolic functions for improved healthspan. A well-designed, randomized, controlled, crossover, feeding study with clinical and molecular mechanistic endpoints is proposed to provide the most definitive level of evidence logistically possible in humans and to establish the role of minimally processed lean pork in healthspan promotion. Utilizing an all-food-provided (dine-in and take-out) design over 18 weeks (rolling recruitment, 8+8, 2w washout), a comprehensive assessment of metabolomics, system biology, physical, and physiological markers that indicate the risk of age-related comorbidities-critical micronutrient deficiency, frailty, metabolic dysfunctions, and cognitive decline, is proposed in upper Midwesterners 65 years and older. A minimally processed plant-forward diet with or without added pork will be compared for over 250 outcome measures using mixed-effects modeling adjusting for covariates in R. n=15/diet/arm i.e., a total starting sample size of n=30 is proposed for 90% power.

ELIGIBILITY:
Inclusion Criteria:

* Generally good health status based on one routine physical in the past 15 months
* Normal HbA1C, weigh 110 lb or more
* Age 65 years or more, generally healthy, all races and both sexes
* Generally practicing a meat-based dietary pattern, do not have any special dietary requirement
* Willingness to comply with the study protocol, including on-site meal consumption and sample/data collection.
* Willing to consume pork as sole meat source during the feeding study.

Exclusion Criteria:

* Tobacco/drug/alcohol use
* Not on any special diet within 3 months of recruitment, and do not have any intention to lose weight.
* Active history of cancer, diabetes, heart, liver, and kidney diseases
* major gastrointestinal disorders in the past 3 months
* history of heart attacks or stroke
* Unable to meet in-person visit requirements for dining, picking up meals, and tests
* Any mental health condition that would affect the ability to provide written informed consent.
* If they were unwilling to abstain from taking certain nutritional supplements, alcohol, or non-study foods during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of Fasting insulin in blood | Time frame: 16 weeks
  Using Microplate assay
Concentration of Ferritin in blood | Time frame: 16 weeks
  Using Microplate assay
Concentration of Homocysteine in blood | Time frame: 16 weeks
  Using Microplate assay
Frequency of Sit-to-stand for strength assessment | Time frame: 16 weeks
  Functional assessment test

SECONDARY OUTCOMES:
Fasting blood glucose concentration in blood | Time frame: 16 weeks
  Using Glucometer
Concentration of FGF21 in blood | Time frame: 16 weeks
  Using Microplate assay
HOMA-IR index using insulin and glucose concentration in blood | Time frame: 16 weeks
  Standard equation
Concentration of ApoB in blood | Time frame: 16 weeks
  Using Microplate assay
Concentration of Lipid panel in blood | Time frame: 16 weeks
  Cholestech ldx
Concentration of IGF-1 in blood | Time frame: 16 weeks
  Using Microplate assay
Concentration of Complex lipids panel in blood | Time frame: 16 weeks
  Using LC/MS based assay
Concentration of C-peptide | Time frame: 16 weeks
  Using Microplate assay
Concentration of HsCRP in blood | Time frame: 16 weeks
  Using Microplate assay
Height in cm | Time frame: 16 weeks
  Measurements
Body Weight in kg | Time frame:16 weeks
  Measurements
Blood pressure in mm Hg | Time frame: 16 weeks
  Upper arm cuff
heart rate in beats per minute | Time frame: 16 weeks
  Upper arm cuff
Grip force per kg mass | Time frame: 16 weeks
  Using Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Moul Dey, Ph.D., Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Wagner Hall 416, Brookings, South Dakota, United States

REFERENCES:
- [Derived] Vaezi S, de Vargas BO, Weidauer L, Freeling JL, Dey M. Effects of Minimally Processed Red Meat within a Plant-Forward Diet on Biomarkers of Physical and Cognitive Aging: A Randomized Controlled Crossover Feeding Trial. Curr Dev Nutr. 2025 Dec 10;10(1):107615. doi: 10.1016/j.cdnut.2025.107615. eCollection 2026 Jan. PMID 41551721
- [Derived] Vaezi S, Freeling JL, de Vargas BO, Weidauer L, Shoemaker ME, Sanders WM, Dey M. Impacts of minimally-processed omnivorous vs lacto-ovo-vegetarian diets on insulin sensitivity, lipid profile, and adiposity in older adults: Secondary findings from a randomized crossover feeding trial. Clin Nutr. 2025 Dec;55:90-103. doi: 10.1016/j.clnu.2025.10.010. Epub 2025 Oct 29. PMID 41202666
- [Derived] Vaezi S, de Vargas BO, Freeling JL, Weidauer L, Dey M. Effects of Minimally Processed Red Meat Within a Plant-Forward Diet on Biomarkers of Physical and Cognitive Aging: A Randomized Controlled Crossover Feeding Trial. medRxiv [Preprint]. 2025 Aug 13:2025.08.11.25333443. doi: 10.1101/2025.08.11.25333443. PMID 40832369
- [Derived] de Vargas BO, Vaezi S, Freeling JL, Zhang Y, Weidauer L, Lee CL, Zhao J, Dey M. Design and Implementation of the Protein-Distinct Macronutrient-Equivalent Diet (PRODMED) Study: An Eighteen-Week Randomized Crossover Feeding Trial Among Free-Living Rural Older Adults. Curr Dev Nutr. 2025 Mar 24;9(5):104588. doi: 10.1016/j.cdnut.2025.104588. eCollection 2025 May. PMID 40291832